CLINICAL TRIAL: NCT02879838
Title: Occupational Respiratory Allergies and Gene-environment Interactions
Acronym: ARPEIGE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: ANSES-2013/ARPEIGE-PENVEN/MS
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Work Related Asthma
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample for collection of human biological material for genotyping analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Occupational Asthma
  Interventions: Other: Blood sample
- Work Aggravated Asthma
  Interventions: Other: Blood sample
- Non-Work-Related Asthma
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Biobank. Analysis of cytokines and DNA polymorphisms

SUMMARY:
The purpose is to compare clinical, functional, professional and socio-economical characteristics of patients with occupational asthma and work aggravated asthma.

Secondary purposes are:

* to evaluate diagnostic value of new non-invasive techniques such as exhaled nitric oxide and cytology of induced expectoration;
* to estimate medical-social becoming of diagnosed work-related asthma after one year;
* to establish a biobank of blood samples of individuals with work related asthma for measurement of cytokines and search for genetic polymorphisms associated with asthma.

DETAILED DESCRIPTION:
Participants with work related asthma or suspected work related asthma will obtain a precise diagnosis concerning severity and control of respiratory disorder and also the possible effect of professional environment on the disorder. Their medical care and medico-legal care, in case of recognition of occupational disease, could be ameliorated.

In general, this study will allow the harmonization of diagnostic care and medical, medico-professional and medico-legal management of cases of work related asthma in specialized hospitals.

ELIGIBILITY:
Inclusion Criteria:

- Patient consulting for suspected work-related asthma in one of hospitals participating to the study

Exclusion Criteria:

* Patient refusing to participate
* Pregnant or breastfeeding women
* Individual in life-threatening emergency
* Hospitalized patient
* Patient in a health or social institution
* Person deprived of liberty
* Person with total occupational disability
* Retired person
* Person diagnosed as non-asthmatic
* Asthmatic person already enrolled in a clinical trial of bio-therapy to treat asthma

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men or women, professionally active, consulting in one of hospitals participating to the study for suspicion of work-related asthma .
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Classification of suspected work-related asthma in occupational asthma, work aggravated asthma, non-work-related asthma | Inclusion
  Interpretation of diagnostic algorithm of study

SECONDARY OUTCOMES:
Nitric oxide level | Inclusion
  Bronchial inflammation marker
Cytology of induced expectoration | Inclusion
  Bronchial inflammation marker
Nonspecific bronchial hyperreactivity evaluated with metacholine bronchial challenge test and/or isocapnic hyperventilation test | Inclusion
Control of asthma symptoms evaluated with Asthma Control test and peak exploratory flow | Inclusion
Severity of symptoms | Inclusion
Costs of different types of asthma | Inclusion and after 1 year
  Direct and induced costs

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Paris, Principal Investigator — Centre de Consultation de Pathologies Professionnelles, CHRU Nancy
Locations (12):
- France (12):
  - Centre de consultation de pathologies professionnelles, Hôpital Pellegrin - CHU de Bordeaux, Bordeaux
  - Centre de consultation de pathologies professionnelles, Hôpital côte de Nacre - CHU de Caen, Caen
  - Centre de consultation de pathologies professionnelles, Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre de consultation de pathologies professionnelles, Hôpital Michallon - CHU de Grenoble, Grenoble
  - Centre de consultation de pathologies professionnelles, immeuble Tourville - CHU de Nantes, Nantes
  - Centre de consultation de pathologies professionnelles, AP-HP groupe hospitalier Cochin, Paris
  - Centre de consultation de pathologies professionnelles, Hôpital Fernand-Widal, Paris
  - Centre de consultation de pathologies professionnelles, Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre de consultation de pathologies professionnelles, Hôpital Civil - CHU de Strasbourg, Strasbourg
  - Centre de consultation de pathologies professionnelles, Hôpital Lyautey - CHU de Strasbourg, Strasbourg
  - Centre de consultation de pathologies professionnelles, Hôpital Purpan - CHU de Toulouse, Toulouse
  - Centre de consultation de pathologies professionnelles, CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No